CLINICAL TRIAL: NCT06771050
Title: The RandOmised Arthroplasty Infection worlDwide Multidomain Adaptive Platform (ROADMAP) Trial
Brief Title: Randomised Arthroplasty Infection Worldwide Multidomain Adaptive Platform (ROADMAP) Trial
Acronym: ROADMAP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Newcastle, Australia (Other)
Collaborators: Hunter Medical Research Institute (HMRI) (Unknown); The University of Western Australia (Other); Michael Garron Hospital (Other); Aotearoa Clinical Trials (Unknown); Exeter Orthopaedic Trial unit (Unknown); University of Sydney (Other); University of Melbourne (Other); The Peter Doherty Institute for Infection and Immunity (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R-2024-0041; 2024015- G2200907 (Other Grant/Funding Number: National Health and Medical Research Council (Australia)); 24/395 (Other Grant/Funding Number: Health Research Council (New Zealand))
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Prosthetic Joint Infections of Hip; Prosthetic Joint Infections of Knee; Large Joint Prosthetic Joint Infections
Keywords: Prosthesis; artificial joint; joint infection; revision; DAIR; Antibiotics; Registry
MeSH Terms: interventions — Debridement

STUDY DESIGN:
Intervention Model Description: Investigator initiated, Randomised Embedded Multifactorial Adaptive Platform (REMAP) trial, conducted across multiple hospitals in several regions of the world.
  ROADMAP is a comparative effectiveness trial comparing two different standard therapy arms with pragmatic approach to treatment randomisation and treatment choices by treating teams. Participants enrolled in the study have the option of deciding whether to be randomised in one or more (if available) treatment domains concurrently, if they meet the eligibility criteria.
  Current domains:
  * Surgical strategy domain
  * Antibiotic duration domain
  * Antibiotic choice domain
  * Other domains to be determined
  The ROADMAP trial will repeatedly fit Bayesian hierarchical logistic models to the accumulating data (interim analyses), over the life of the trial, to estimate model parameters and evaluate pre-specified decision criteria either within a cell or a whole domain.
Masking Description: This will be an open-label study unless otherwise specified in a domain-specific appendix. For the overall data and results, only specified members of the statistical analytical team and Data and Safety Monitoring Committee (DSMC) will have access to unblinded results, with other trial investigators and staff remaining blinded to the aggregate results until completion of final analysis for a domain or cell.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1. SURGICAL DOMAIN: Late Acute Silo (Active Comparator): Surgical Domain comparing outcomes of surgical strategies - Debridement and implant retention (DAIR) versus Revision arthroplasty (either one stage or two stage at the discretion of the treating surgeon)
  Interventions: Procedure: Debridement and Implant Retention (DAIR)
- 2. ANTIBIOTIC CHOICE DOMAIN (Active Comparator): Backbone therapy alone (active comparator) versus Backbone antibiotic therapy plus Rifampicin.
  Interventions: Drug: Antibiotic Choice
- 3. ANTIBIOTIC DURATION DOMAIN Part A - Single Stage Revision (Active Comparator): Length of antibiotic course duration after a single stage revision, short course (6 weeks) versus long course (12 weeks).
  Interventions: Drug: Antibiotic duration Part A - Single stage revision
- 4. ANTIBIOTIC DURATION DOMAIN Part B - Two Stage Revision (Active Comparator): No extended antibiotic prophylaxis versus extended antibiotic prophylaxis following a two-stage revision.
  Interventions: Drug: Antibiotic Duration Part B - Two stage revision

INTERVENTIONS:
Procedure: Debridement and Implant Retention (DAIR) — Intervention 1: DAIR- cleaning of infected joint including irrigation, debridement and exchange of modular components (those not fixed to bone) with implant retention.
  Intervention 2: Single stage revision - cleaning of infected joint including irrigation, removal and placement of "definitive" new components which could be primary or revision components.
  Other Names: Revision Arthroplasty - Single stage revision
  Arms: 1. SURGICAL DOMAIN: Late Acute Silo
Drug: Antibiotic Choice — No intervention: Backbone antibiotic therapy only depends on the organism and is detailed in the protocol.
  Intervention: Backbone antibiotic therapy plus rifampicin. Dosage 600-900mg per day orally for as long as oral antibiotic treatment continues, but not more than 12 weeks. Prescribed according to local recommended practices and dosed as per local therapeutic guidelines.
  Other Names: No intervention: Standard of Care "Backbone antibiotics"; Intervention: Standard of care " Backbone antibiotics" + Rifampicin antibiotics
  Arms: 2. ANTIBIOTIC CHOICE DOMAIN
Drug: Antibiotic duration Part A - Single stage revision — Intervention Arm: Short course 6-week (42 +/- 7 days) antibiotic course - combined intravenous and oral with antibiotic choice according to organism and patient tolerability factors.
  Intervention Arm: Long course 12- week (84 +/- 7 days) antibiotic course - combined intravenous and oral with antibiotic choice according to organism and patient tolerability factors.
  Other Names: shorter duration - 6 weeks; longer duration - 12 weeks
  Arms: 3. ANTIBIOTIC DURATION DOMAIN Part A - Single Stage Revision
Drug: Antibiotic Duration Part B - Two stage revision — Intervention Arm: Extended prophylaxis for 12 weeks after the 2nd stage revision surgery.
  Intervention Arm: No extended antibiotic prophylaxis after the 2nd stage revision surgery.
  Antibiotic choice by treating team with reference to the original causative organism(s), susceptibility and patient tolerability.
  Other Names: Extended antibiotic prophylaxis following 2nd stage Revision operation; No extended antibiotic prophylaxis following 2nd stage Revision operation
  Arms: 4. ANTIBIOTIC DURATION DOMAIN Part B - Two Stage Revision

SUMMARY:
Artificial joint infections are treated with different types of antibiotics and surgery. The ROADMAP study aims to find out which treatments currently used work best in regards to surgery, antibiotic choice as well as the time taking antibiotics. The study will compare different treatments against each other to see which treatment or treatment combination works to provide the best outcome and cure at 12 months. The study will focus on adults with infected artificial hips and knees.

ROADMAP trial looks at normal good clinical care and does not ask any person taking part in the study to have any extra tests or treatments.

If a person takes part in the study they will:

* Sign a consent form
* Give permission for infection and treatment information to be collected and entered into a central ROADMAP specific database and a separate registry of prosthetic joint infection patients. This medical information will include participants medical history, test results and treatment they received. The study will also collect information about medical care and how the participant is feeling at Day 100 and Day 365 (1 year) after starting the study.

There are several different study parts. Each part focuses on research focus areas called domains. ROADMAP has 3 different domains; 1. Surgical, 2. Antibiotic choice and 3. Antibiotic Duration domains. Not every hospital is taking part in all 3 domains and if someone chooses to participate they do not have to participate in all domains. Specific domain details are:

1. Surgical Treatment Domain This domain will find out if it is better to do an operation to clean out the infection but keep the artificial joint in place (this is called a Debridement, Antibiotics and Implant Retention operation (DAIR)) or to clean out the infection and swap the artificial joint out for a new one (this is called a "revision" operation).

   DAIR usually involves a single operation but sometimes needs more. Revision surgery may be done in one operation (single stage revision) or two operations (two stage revision). Previous research has suggested that cure rates may be better with revision operations than with DAIR, but this is not clear.

   If the participant consents to the surgical domain they will be randomly allocated to either a DAIR, to clean the artificial joint but keep it in place, or to have surgery that cleans and replaces the artificial joint with a new one (revision). A revision operation, may involve one (single stage) or two different surgeries which can be days, weeks or months apart (two stage).

   The participants surgeon and treating team in consultation with the participant will decide what kind of treatment they are best to receive, DAIR, single stage or two stage revision.
2. Antibiotic Choice Domain Many different microorganisms (germs) can cause artificial joint infections and many different antibiotics are used to fight infections. ROADMAP will look at different antibiotics commonly used to treat artificial joint infection. This domain will focus on an antibiotic called rifampicin (also sometimes known as rifampin) as it is often added to other antibiotics to help treat artificial joint infections. Rifampicin is not a new antibiotic but it is not clear if treatment cure rates are better if it is added.

   All people taking part in this domain will be given antibiotics that will treat their artificial joint infection, called the "backbone antibiotics", but some will be given "backbone antibiotics" plus rifampicin. "Backbone antibiotics" can be either one antibiotic or a number of different antibiotics. These will be given into a vein (IV) at first, and will be changed to tablets or capsules later.

   All antibiotics in this domain are commonly used and the "backbone antibiotics" will be chosen by treating doctors after looking at the type of germ and what antibiotic may work for the germ, as well as medical history including past antibiotic reactions. Antibiotics are taken for approximately 12 weeks after DAIR surgery, however after revision surgery then the time taking antibiotics may be shorter or longer.
3. Antibiotic Duration Domain Antibiotic treatment times are the focus of this domain as it is not clear how long someone should take antibiotics when revision surgery is used to treat artificial joint infection. To show what antibiotic time period is best for treatment and cure people who have had revision surgery participating in this domain will receive either "standard" or "extended" duration of antibiotics.

In this domain, after a one-stage revision, the participant will be randomised to have either 6 weeks or 12 weeks of antibiotics after the operation. If a two-stage revision operation has been done the participant will receive around 6 weeks of antibiotics between the two operation stages. After the two stage revision has been completed the participant will be randomised to either stop antibiotics or have a further 12 weeks of antibiotic treatment.

DETAILED DESCRIPTION:
Over 120,000 hip or knee replacements are performed in Australia every year, and there are ~1 million Australians living with one or more joint replacements. Approximately 3,900 prosthetic joint infections (PJI) are diagnosed in Australia every year. The burden is similar in other resource-rich countries. For example, in Canada, over 130,000 hip and knee replacements are performed yearly and 2% of primary arthroplasties require a revision within 2 years. Infection has been identified as the most common cause for a revision surgery, which translates to $42.1 million CAD in inpatient costs to the Canadian health care system.

PJIs are difficult to treat, because of the presence of a foreign body, which encourages biofilm formation, and the need for combined surgical and prolonged antibiotic management. Outcomes are generally poor, with substantial variation in reported treatment success (ranging from 10 to 90%, median 50% after 2 years) and PJIs have striking health care costs. Existing treatment guidelines are informed by low quality evidence, with fewer than 1,700 participants ever enrolled into published randomised controlled trials comparing management approaches. Defining the optimal surgical and antibiotic approaches to PJI is a critical unmet need.

The Investigators are using an adaptive platform trial to allow the investigators to simultaneously address these questions in the management of PJI. The trial will include 3 silos (Early, Late Acute and Chronic PJI) and evaluate treatments and outcome of treatments over a 12 month period. Time points for data collection and analysis will be Day 100 and Day 365 post platform entry.

The Investigators plan to test interventions within 3 initial domains of:

1. Surgical Domain comparing outcomes of surgical strategies - Debridement and Implant Retention (DAIR) vs Revision arthroplasty.
2. Antibiotic Choice Domain comparing outcomes of antibiotic treatment - Backbone antibiotic regimen plus the addition of oral rifampicin (AKA rifampin) vs Backbone antibiotic regimen without rifampicin.
3. Antibiotic Duration Domains comparing the duration of antibiotics treatment in relation to one stage and also two stage surgical Revision arthroplasty strategies

   1. Part A - PJI treatment with a single-stage revision - 6 weeks (+/-7 days) of antibiotics following the single stage revision procedure ('short course regimen') vs 12 weeks (+/-7 days) of antibiotics following the single stage revision procedure ('long course regimen')
   2. Part B - PJI treatment with a two-stage revision and negative cultures following reimplantation (second stage) - Extended antibiotic prophylaxis: 12 weeks vs No extended prophylaxis.

The ROADMAP trial infrastructure will also have the potential to add further domains to the platform.

RANDOMISATION Participants will be randomly allocated to one arm within each domain for which they are eligible, which their site is participating in, and for which they have consented, using a web-based module available 24h a day 7 days a week. Randomisation within the patient's known silo, for all available domains will occur immediately following provision of consent (which is considered the time of platform entry), however, the reveal of each treatment allocation(s) will be delayed subject to confirmation of domain eligibility.

BLINDING This will be an open-label study unless otherwise specified in a domain-specific appendix. For the overall data and results, only specified members of the statistical analytical team and Data and Safety Monitoring Committee (DSMC) will have access to unblinded results, with other trial investigators and staff remaining blinded to the aggregate results until completion of final analysis for a domain or cell.

ANALYSIS The ROADMAP trial will repeatedly fit Bayesian hierarchical logistic models to the accumulating data (interim analyses), over the life of the trial, to estimate model parameters and evaluate pre-specified decision criteria either within a cell or a whole domain.

CORE PRIMARY OUTCOME MEASURE Treatment success assessed at 12 months post-platform entry, defined as all of: i) Alive; ii) Clinical cure (no clinical or microbiological evidence of infection); iii) No ongoing use of antibiotics for the index joint; and iv) "Destination prosthesis" (the prosthesis present after the initial management strategy is complete) still in place

CORE SECONDARY OUTCOME MEASURES

A core set of secondary endpoints will be evaluated across all domains:

1. A "desirability of outcome ranking" (DOOR - an ordinal outcome which ranks participants based on a combination of clinical cure, patient-reported joint function and quality of life).
2. Patient-reported joint function (Oxford hip or knee score) at 12 months after platform entry.
3. Patient-reported quality of life (EQ5D5L) at 12 months after platform entry
4. Cost effectiveness
5. All-cause mortality at 12 months after platform entry
6. "Clinical cure" at 12 months after platform entry
7. Proportion alive and no longer taking any antibiotics for the index joint at 12 months after platform entry.
8. Proportion in whom the destination prosthesis is still in place at 12 months after platform entry.
9. Microbiological relapse (Positive joint fluid or tissue culture for one or more of the index isolates between Day 100 and 12 months after platform entry)
10. Microbiological reinfection (Positive joint fluid or tissue culture with a different organism to all of the index isolates between Day 100 and 12 months after platform entry).
11. Time alive and free from any revision procedure on the index joint captured by a national joint replacement registry within 24 months of platform entry

ROADMAP Registry ROADMAP registry is a planned adjunct to the ROADMAP main platform study. The ROADMAP registry aims to describe the entire group of people who get large joint prosthetic joint infections, many of whom have never been a part of other previous research studies. The ROADMAP registry is interested in the different factors that can be examine to identify patterns in the medical history of people that get prosthetic joint infections, what sorts of testing and treatments they receive, and how these might affect their outcome. The registry information when analysed will be used to improve knowledge about prosthetic joint infections and also patient care.

The registry will include participants of the main platform study and also seek independent consent from patients with prosthetic joint infection that choose not to participate in the main platform study. Data for the registry will be collected from participants medical records with participant provided permissions. In addition, all ROADMAP registry participants will be asked to provide specific consent for data linkage that may occur with existing datasets, such as hospital records, national joint replacement registries, and registries of birth, deaths and marriages.

Apart from collecting available information from medical records, there are no additional tests or treatments involved.

ELIGIBILITY:
Inclusion Criteria:

1. "Confirmed" or "Likely" Prosthetic joint infection of a large joint according to European Bone and Joint Infection Society (EBJIS) criteria (2021)
2. Physically present at participating hospital at time of eligibility assessment
3. "Current" prosthetic joint infection, meaning symptoms and/or signs of the PJI are present at the time of eligibility assessment.

Exclusion Criteria:

Potentially eligible participants meeting any of the following criteria at the time of eligibility assessment for platform entry will be excluded from the randomised platform (but may still participate in the registry):

1. The index prosthetic joint is a shoulder, elbow, wrist or ankle.
2. Known previous participation in the randomised ROADMAP randomised platform for the index joint.
3. Known previous participation in the randomised ROADMAP platform for a joint other than the index joint within the 12 months prior to eligibility assessment
4. Treating clinician believes that death is imminent and inevitable.
5. Treatment is not with curative intent.
6. Patient is not classifiable into one of the three defined silos.
7. Patient is unlikely to be accessible for follow up over the 12 months following platform entry.
8. Treating team deems enrolment in the study is not in the best interests of the patient.

To be included in any of the following Domains the participant must be eligible for the PLATFORM ( as listed above) and none of the platform-level exclusion criteria AND all of the domain-level inclusion and none of the domain-level exclusion criteria.

Domain-specific eligibility criteria Each domain may have additional criteria for eligibility. Participants who fulfil the above criteria will be assessed for enrolment into all domains active at a participating site. At least 2 interventions (which may include standard of care) within a domain must be available to an eligible participant in order for that participant to enter the domain. The minimum number of interventions within a domain is two. The availability of interventions within domains will be region- and site-specific, although the default position is that all interventions within a domain will be available at all sites.

Surgical Strategy Domain: Late Acute Silo inclusion criteria

Patient is in the Late Acute silo, meaning all of the following 3 criteria are met:

1. Onset of symptoms is >30 days after implantation of the index joint
2. Treating team feel that either DAIR or revision is appropriate for this patient.
3. The infected prosthesis is a primary arthroplasty. Surgical Strategy Domain: Late Acute Silo exclusion criteria

<!-- -->

1. Any previous episode of native joint septic arthritis or PJI in the index joint
2. A definitive DAIR has already occurred for this episode of infection.
3. A revision has already occurred for this episode of infection
4. Loosening or instability of any component of the prosthesis
5. Predicted inadequate soft tissue coverage for wound closure
6. One or more of the causative organisms is a fungus or a "difficult to treat" bacterium.
7. Treating team deems enrolment in this domain is not in the best interests of the patient.

Antibiotic Choice Domain inclusion criteria

1. The time of eligibility assessment is between 48h and 7 days following initial surgical treatment.
2. One or more of the causative organisms is a Gram-positive of interest OR the infection is culture negative.

   Antibiotic Choice Domain exclusion criteria

<!-- -->

1. Previous hypersensitivity reaction to rifampicin
2. The patient is receiving a concomitant medication with an expected clinically significant drug interaction with rifampicin, which cannot be ceased, substituted for an alternative agent, or mitigated by dose adjustment.
3. One or more causative Gram-positive organisms of interest have in-vitro evidence of resistance to rifampicin
4. Known pregnancy or breastfeeding
5. Treating team deems enrolment in this domain is not in the best interests of the patient.

Antibiotic Duration Part A Domain inclusion criteria

1. A single stage revision procedure has been performed

   For the purposes of this domain, the definition of a single stage revision procedure is as follows:

   A one-stage revision means:

   • Arthrotomy

   • Removal of all prosthetic components

   • Comprehensive synovectomy

   • Placement of "definitive" new components
   * could be primary or revision components • With no plans for a second stage operation

   Additional recommended elements (not part of definition, but considered 'ideal' elements of this procedure):
   * Removal of all loose cement; well-fixed cement may be retained.
   * Double set up (using a separate set of sterile instruments and drapes for the reimplantation)

   Antibiotic Duration Part A Domain exclusion criteria

   Patients will be excluded from this domain if, at the time of eligibility assessment, they have any of the following:

<!-- -->

1. Any causative organism is a fungus or a 'difficult-to-treat' bacterium at the time of platform entry
2. Treating team deems enrolment in this domain is not in the best interests of the patient
3. The single stage revision was >7 days ago
4. Patient no longer willing to participate in the domain

Antibiotic Duration Part B Domain Eligibility assessment and allocation reveal will be performed at day 7 (+/- 3 days) from the time of the reimplantation operation - i.e. between 4 and 10 days following the reimplantation operation. The purpose of this time frame is to confirmation of negative reimplantation cultures.

Antibiotic Duration Part B Domain inclusion criteria

1. A two-stage revision procedure has been performed

   For the purposes of this domain, the definition of two-stage revision and reimplantation procedures are defined as follows:

   A two-stage revision means:

   • Removal of all existing prosthetic components (including metal, ceramic, polyethylene) and any loose cement
   * Placement of a temporary prosthesis or spacer with the intention to replace this at a later time point with a permanent prosthesis
   * The intention to subsequently replace of the temporary spacer with a definitive prosthesis at a reimplantation operation in the future

   Additional recommended elements (not part of definition, but encouraged):

   • Use of antibiotic-loaded cement as the spacer
   * Use of an articulating spacer which is capable of withstanding weight-bearing

   A reimplantation procedure as the second stage of a two-stage revision means:

   • Removal of the temporary prosthesis and all associated cement
   * Implantation of a new prosthesis; considered the 'destination prosthesis'
2. The infected prosthesis was a primary (not revision) arthroplasty
3. At least 6 weeks of antibiotics have been received following the first stage revision, intended as treatment of the index infection
4. The reimplantation operation was done 4-10 days ago

Antibiotic Duration Part B Domain exclusion criteria

1. >6 months has passed since platform entry
2. One or more of the causative organisms is a fungus or a 'difficult-to-treat' bacterium
3. No perioperative tissue or fluid cultures were collected at the reimplantation operation
4. Perioperative cultures collected at reimplantation grow a significant organism (s)
5. Long-term antibiotic suppressive therapy is planned following the reimplantation operation
6. Treating team deems enrolment in this domain is not in the best interests of the patient
7. Patient no longer willing to participate in the domain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2025-03-26 (Estimated); Primary Completion 2028-02-18 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment success at 12 months | up to 13 months (with a window of up to 13 months i.e. 365 to 395 days) after platform entry.
  The primary endpoint for all cells and domains will be treatment success at 12 months, defined as ALL FOUR OF: 1. Patient is alive. 2. Clinical cure = no clinical or microbiological evidence of ongoing infection in the index joint 3. The patient is no longer taking antibiotics for the index joint. 4. The destination prosthesis is still in place. The primary endpoint is determined through a search of hospital databases for a record of participant's death, or follow-up contact with participant's community healthcare provider, or follow-up contact with patient or their nominated carer, or linkage with death registries. The preferred method is through direct face to face clinic visit. However, phone contact with the patient may occur. In addition, any or all of the four components of the primary endpoint can be derived from external data such as GP records or specialist letters.

SECONDARY OUTCOMES:
A "desirability of outcome ranking" DOOR | Platform entry until day 265
  DOOR - A "desirability of outcome ranking" Each element of this composite ordinal outcome (DOOR) is already included as an endpoint in its own right (clinical cure, mortality, Oxford joint score and EQ5D5L). The DOOR is simply a way of using a combination of these outcomes to rank participants and then compare the ranks between two treatments. DOOR - an ordinal outcome which ranks participants based on a combination of the endpoints A: Clinical Cure - Primary outcome measure 1. B: Mortality - Primary outcome measure 1. C: Oxford Joint Score - Secondary outcome 3. D: EQ5D5L - Secondary outcome 4.
Patient-reported joint function (Oxford hip or knee score) at 12 months after platform entry. | platform entry until day 365
  Log cumulative odds ratio of intervention compared to domain control for having Oxford hip or knee score j or higher compared to j-1 or lower (assumed constant for all j), within a domain (d) and estimated for each silo (s)
Patient-reported quality of life (EuroQol-5 Dimensions-5 Levels (EQ5D5L)) at 12 months after platform entry. | Platform entry until day 365
  Difference in mean EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) utility score between intervention and control group within a domain (d) and estimated for each silo (s).ED-5D-5L consists of EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Cost effectiveness over the first 12 months after platform entry. | From platform entry until day 365
  Bayesian statistical techniques - Monte Carlo simulation-used to estimate incremental cost-effectiveness ratios and net monetary benefits for each treatment comparison. Incremental costs and outcomes are measured arithmetic mean differences with prior distributions informed by observed data. Resource use data over 12 month follow up period.; 1)treatment costs 2) surgical cost including implant costs 3) operating theatre costs 3) ICU lengths of stay, and 4) readmissions. Quality-adjusted life years calculated using EQ-5D-5L at baseline and 12 months. To incorporate data uncertainty, results will be reported using mean of 10,000 simulations, alongside 95% credible intervals. Overall results will be presented as a probability of an intervention being cost-effective, which has the advantage of being easily interpreted. Deterministic (one-way) and probabilistic sensitivity analyses to test assumptions in modelling and impact of changing key parameters, and joint parameter uncertainty.
All-cause mortality at 12 months after platform entry | From platform entry until day 365
  Determined through hospital database search for record of participant death, or follow-up contact with the participant's community care provider, or with the patient or their nominated carer, or linkage with death registries. Log odds ratio of all-cause mortality at 12 months between intervention and control groups within a domain (d), estimated for each silo (s).
"Clinical cure" at 12 months after platform entry (as defined in the primary outcome) | From platform entry until day 365
  Clinical cure = no clinical or microbiological evidence of ongoing infection in the index joint. Clinical evidence includes any of local redness and tenderness, joint effusion, a draining sinus, or wound breakdown. Microbiological evidence includes positive cultures of synovial fluid or periprosthetic tissue of one or more of original index causative organism(s). Log odds ratio of clinical cure between intervention and control groups within a domain (d), estimated for each silo (s).
Proportion alive and no longer taking any antibiotics for the index joint at 12 months after platform entry (as defined in the primary outcome). | From platform entry until day 365
  To be considered "not taking antibiotics", the patient should not have received any antibiotics for the index joint for at least the past 6 weeks (42 days). Log odds ratio of the patient no longer taking any antibiotics for the index joint between intervention and control groups within a domain (d), estimated for each silo (s).
Proportion in whom the destination prosthesis is still in place at 12 months after platform entry (as defined in the primary outcome) | From platform entry until day 365
  Log odds ratio of the destination prosthesis still being in place between intervention and control groups within a domain (d), estimated for each silo (s).
Microbiological relapse | From platform entry until day 100 and day 365
  (Positive joint fluid or tissue culture of the same genus and species as one or more of the index isolates between 100 days and 12 months after platform entry). The index isolate(s) are defined as all organisms identified from specimens collected between the date of diagnosis and 10 days post platform entry, which are judged as clinically significant causative organisms by the treating team and site PI. Log odds ratio of treatment success between intervention and control groups within a domain (d), estimated for each silo (s).
Microbiological reinfection | From platform entry until day 100 and day 365
  (Positive joint fluid or tissue culture with a different organism to any of the index isolates between 100 days and 12 months after platform entry). Log odds ratio of treatment success between intervention and control groups within a domain (d), estimated for each silo (s)
Time alive and free from any revision procedure on the index joint captured by a national joint replacement registry within 24 months of platform entry | From platform entry until 24 months
  Median difference in time to revision procedure or death between intervention and control groups within each domain. Note this endpoint will only be available for the subset of patients who have data linked to a national joint registry.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua S Davis. Co-chief Investigator, infectious diseases Specialist, Study Director — University of Newcastle, Menzies Institute, Hunter Medical Research Institute, Hunter New England Health; Laurens Manning, Co-chief Investigator, infectious diseases Specialist, Study Director — The University of Western Australia
Locations (31):
- Australia (31):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Mater Hospital Sydney ST Vincents Network, North Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Prince Charles Hospital, Chermside, Queensland
  - Townsville Hospital and Health Service, Douglas, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Calvary Adelaide Private Hospital, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Eastern Health, Box Hill, Victoria
  - Epworth Hospital, Box Hill, Victoria
  - Dandenong/Monash Hospital, Dandenong, Victoria
  - Northern health, Epping, Victoria
  - St Vincents, Fitzroy, Victoria
  - Western Health, Footscray, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Fiona Stanley Hospital, Murdoch, Western AustraliaA

IPD SHARING:
Plan to Share IPD: No
Study data can be requested for future research through contacting the study team and requesting access. The Global Clinical Trial Management Team will review applications and approve or decline applications based on researcher supplied information. The ROADMAP trial Has in development a Publication policy and also a data access policy which protects the data prior to publication in open sources.